CLINICAL TRIAL: NCT05597150
Title: To Explore the Regulatory Effect of Magnesium on Intestinal Flora in Healthy Adults # A Single-center, Prospective, Self-controlled Trial
Brief Title: The Exploration of the Regulatory Effect of Magnesium on Intestinal Flora in Healthy Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Seventh Affiliated Hospital, Southern Medical University (Other)
Responsible Party: Principal Investigator, Yu Chen, chief physician, The Seventh Affiliated Hospital, Southern Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: (2022)--0009
Record Dates: First submitted 2022-10-24; First posted 2022-10-27 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Healthy State
Keywords: magnesium, gut microbiota, healthy adult
MeSH Terms: interventions — magnesium citrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental Group (Experimental)
  Interventions: Dietary Supplement: Magnesium Citrate

INTERVENTIONS:
Dietary Supplement: Magnesium Citrate — Each participant should receive a high-magnesium diet for 1-3 weeks and take magnesium supplements for 4-6 weeks.

SUMMARY:
In this A Single-center, Prospective, Self-controlled trial, subjects should avoid a high-magnesium diet for 1-3 weeks and take magnesium supplements for 4-6 weeks.

DETAILED DESCRIPTION:
Investigational drug# Oral magnesium Study title# To explore the regulatory effect of magnesium on intestinal flora in healthy adults # A Single-center, Prospective, Self-controlled trial.

Principal Investigator# Professor Yu Chen, Department of Gastroenterology, The Seventh Affiliated Hospital, Southern Medical University.

Professor Peng Chen, Department of Pathophysiology, School of Basic Medical Sciences, Southern Medical University.

Study subjects# Healthy adult, Age 20-30 years Study phase# Investigator Initiated Trial(IIT) Study objectives# The objective of the study is to explore the regulatory effect of magnesium on intestinal flora in healthy adults Study design# A Single-center, Prospective, Self-controlled trial. Medication method# Subjects should avoid high magnesium diet for 1-3 weeks, and take magnesium supplement (food grade magnesium citrate: three capsules a day, after meals, 400mg magnesium) in 4-6 weeks. Peripheral blood and stool samples were collected from 60 subjects on day 0, day 21, and day 42 of the study period for routine blood tests, blood biochemical tests, and 16s rDNA sequencing analysis of gut microbiota.

Course#42days Sample size#60.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged 20-30 years in the general community
* Without gender or ethnic requirements, who did not participate in other trials at the same time, volunteered to participate in this study
* No underlying diseases.

Exclusion Criteria:

* (1) Patients who have taken antibiotics orally in the past 3 months or have acute or chronic inflammation;
* (2) Those who have taken hormones within 3 months;
* (3) Those who have taken drugs that may interfere with glucose and lipid metabolism (such as insulin, glyburide, indomethacin, phentolamine, fuuside, phenytoin sodium, cortisone, etc.) and those who have taken probiotics within 1 month;
* (4) smokers and drinkers;
* (5) Uncontrollable mental disorders (including hospitalization history of mental illness);
* (6) Currently attending a weight loss or weight management course;
* (7) prescribed diet for specific or other reasons (e.g. celiac disease);
* (8) pregnant or lactating women;
* (9) Patients with cardiac and renal insufficiency;
* (10) Long-term constipation.

Ages: 20 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2022-10-15 (Actual); Primary Completion 2023-01-30 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
16S rDNA sequencing | 21days, 42 days
  16S rDNA sequencing technology was used to identify the structural and functional changes of intestinal microbiota before and after magnesium supplementation.
Metabolomic analysis of serum and feces | 21days, 42 days
  To determine the alteration of gut microbiota and their metabolites after Mg supplementary.
Number of participantswith abnormal laboratory tests results | 21days, 42 days
  If there are abnormal situations during the experiment that may pose significant risks to the health or safety of the participants, the research team may need to terminate the experiment to ensure participant safety. Only

SECONDARY OUTCOMES:
The plasma levels of Mg2+ in each study phase. | 21days, 42 days
  The plasma levels of Mg2+ would be detected on day 21 and day 42.
Total bilirubin concentration after 21days oral Mg. | 21days, 42 days
  change from 21days in Total bilirubin and analyzed by the AU5800 fully automatic biochemical analyzer.
Direct bilirubin concentration after 21days oral Mg. | 21days, 42 days
  change from 21days in Direct bilirubin and analyzed by the AU5800 fully automatic biochemical analyzer.
Indirect bilirubin concentration after 21days oral Mg. | 21days, 42 days
  change from 21days in indirect bilirubin and analyzed by the AU5800 fully automatic biochemical analyzer.
uric acid concentration after 21days oral Mg. | 21days, 42 days
  change from 21days in uric acid and analyzed by the AU5800 fully automatic biochemical analyzer.
total triglyceride concentration after 21days oral Mg. | 21days, 42 days
  change from 21days in total triglyceride and analyzed by the AU5800 fully automatic biochemical analyzer.
total protein concentration after 21days oral Mg. | 21days, 42 days
  change from 21days in total protein and analyzed by the AU5800 fully automatic biochemical analyzer.
aspartate transaminase concentration after 21days oral Mg. | 21days, 42 days
  change from 21days in aspartate transaminase and analyzed by the AU5800 fully automatic biochemical analyzer.
alanine transaminase concentration after 21days oral Mg. | 21days, 42 days
  change from 21days in alanine transaminase and analyzed by the AU5800 fully automatic biochemical analyzer.
albumin concentration after 21days oral Mg. | 21days, 42 days
  change from 21days in albumin and analyzed by the AU5800 fully automatic biochemical analyzer.
total cholesterol concentration after 21days oral Mg. | 21days, 42 days
  change from 21days in total cholesterol and analyzed by the AU5800 fully automatic biochemical analyzer.
Urea concentration after 21days oral Mg. | 21days, 42 days
  change from 21days in urea and analyzed by the AU5800 fully automatic biochemical analyzer.
HDL-C concentration after 21days oral Mg. | 21days, 42 days
  change from 21days in HDL-C(high density lipoprotein cholesterol) and analyzed by the AU5800 fully automatic biochemical analyzer.
LDL-C concentration after 21days oral Mg. | 21days, 42 days
  change from 21days in LDC-C(low density lipoprotein cholesterol) and analyzed by the AU5800 fully automatic biochemical analyzer.
Red blood cells analysis after 21days oral Mg. | 21days, 42 days
  change from 21days in Red blood cells and determined by a Sysmex-xn-2000 automatic blood cell analyser.
Plateltes analysis after 21days oral Mg. | 21days, 42 days
  change from 21days in Plateltes cells and determined by a Sysmex-xn-2000 automatic blood cell analyser.
Neutrophil cells analysis | 21days, 42 days
  change from 21days in Neutrophil cells and determined by a Sysmex-xn-2000 automatic blood cell analyser.
Eosinophil cells analysis after 21days oral Mg. | 21days, 42 days
  change from 21days in Eosinophil cells and determined by a Sysmex-xn-2000 automatic blood cell analyser.
Basophil cells analysis after 21days oral Mg. | 21days, 42 days
  change from 21days in Basophil cells and determined by a Sysmex-xn-2000 automatic blood cell analyser.
Lymphocyte cells analysis after 21days oral Mg. | 21days, 42 days
  change from 21days in Lymphocyte cells and determined by a Sysmex-xn-2000 automatic blood cell analyser.
Monocyte cells analysis after 21days oral Mg. | 21days, 42 days
  change from 21days in Monocyte cells and determined by a Sysmex-xn-2000 automatic blood cell analyser.
The fecal Mg2+ concentration in each study phase. | 21days, 42 days
  The fecal Mg2+ concentration would be detected on day 21 and day 42.

CONTACTS AND LOCATIONS:
Locations (1):
- Southern Medical Unversity,the seventh affiliated hospita, Foshan, Guangdong, China

IPD SHARING:
Plan to Share IPD: No
since some data may involve subject's privacy #we have no plans to share data so far# and some data may be shared later depending on the subjects's wishes.

REFERENCES:
- [Derived] Li D, Chen Y, Wan M, Mei F, Wang F, Gu P, Zhang X, Wei R, Zeng Y, Zheng H, Chen B, Xiong Q, Xue T, Guan T, Guo J, Tian Y, Zeng LY, Liu Z, Yuan H, Yang L, Liu H, Dai L, Yu Y, Qiu Y, Wu P, Win S, Than TA, Wei R, Schnabl B, Kaplowitz N, Jiang Y, Ma Q, Chen P. Oral magnesium prevents acetaminophen-induced acute liver injury by modulating microbial metabolism. Cell Host Microbe. 2024 Jan 10;32(1):48-62.e9. doi: 10.1016/j.chom.2023.11.006. Epub 2023 Dec 5. PMID 38056458